CLINICAL TRIAL: NCT03540901
Title: Effect of Acetazolamide on Lung Water Content by Ultrasound in Patients With Respiratory Disease at Altitude: A Randomized, Placebo-controlled, Double-blind Parallel Trial
Brief Title: Effect of Acetazolamide on Lung Water Content by Ultrasound in Patients With Respiratory Disease at Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-00137G
Record Dates: First submitted 2018-05-15; First posted 2018-05-30 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: prevention; acetazolamide; obstructive airway disease; lung water
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACETAZOLAMIDE oral capsule (Active Comparator): 375mg/day (capsule @125 mg: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3100m until the morning after the second night at 3100m
  Interventions: Drug: ACETAZOLAMIDE oral capsule
- PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3100m until the morning after the second night at 3100m.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ACETAZOLAMIDE oral capsule — Administration of 125mg acetazolamide in the morning, 250mg in the evening, starting 24 hours before departure to 3100m
  Arms: ACETAZOLAMIDE oral capsule
Drug: Placebo oral capsule — Administration of equally looking placebo capsules in the morning and evening, starting 24 hours before departure to 3100m
  Arms: PLACEBO oral capsule

SUMMARY:
This trial will evaluate the effect of acetazolamide (375 mg per day) vs. placebo on lung water content by ultrasound at acute altitude exposure in patients with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind parallel trial evaluating the effect of acetazolamide (375 mg per day) vs. placebo on lung water content by ultrasound in lowlanders with chronic obstructive pulmonary disease travelling to altitude. Participants living in the Bishkek area, Kyrgyzstan (760m), will be transferred by car within 4h to the Tuja Ashu high altitude clinic (3100 m), and stay there for 2 days. Acetazolamide 375mg/day (or placebo) will be administered 24 hours before departure at 760 m and during the stay at altitude. Outcomes will be assessed during the stay at 3100 m.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age 18-75 yrs.
* COPD diagnosed according to GOLD, FEV1 40-80% predicted, Oxygen Saturation (SpO2) ≥92% at 750 m.
* Born, raised and currently living at low altitude (<800m).
* Written informed consent.

Exclusion Criteria:

* COPD exacerbation, very severe COPD with hypoxemia at low altitude (FEV1/Forced Vital Capacity <0.7, FEV1 <40% predicted, oxygen saturation on room air <92% at 750 m).
* Comorbidities such as uncontrolled cardiovascular disease, i.e., unstable systemic arterial hypertension, coronary artery disease; previous stroke; obstructive sleep apnea; pneumothorax in the last 2 months.
* Internal, neurologic, rheumatologic or psychiatric disease including current heavy smoking (>20 cigarettes per day)
* Known renal failure or allergy to acetazolamide and other sulfonamides

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Difference in change of ultrasound lung comets from 760 m baseline measurement to measurement at 3100 m in the acetazolamide compared to the placebo group | Day 2 at 760m and 3100m
  Difference in change of ultrasound lung comets from 760 m baseline measurement to measurement at 3100 m in the acetazolamide compared to the placebo group

SECONDARY OUTCOMES:
Change of ultrasound lung comets from 760 m baseline measurement to measurement at 3100 m in the acetazolamide and in the placebo group, respectively | Day 2 at 3100m
  Change of ultrasound lung comets from 760 m baseline measurement to measurement at 3100 m in the acetazolamide and in the placebo group, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan; Michael Furian, MSc, Principal Investigator — University Hospital, Zürich; Silvia Ulrich, MD, Principal Investigator — University Hospital, Zürich
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan